CLINICAL TRIAL: NCT02236741
Title: The Use of Pramipexole and Other Dopamine Agonists and the Risks of Heart Failure and Pneumonia
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.672
Record Dates: First submitted 2014-09-10; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- users of anti-parkinsonian drugs
  Interventions: Drug: Mirapexin® (Sifrol®)

INTERVENTIONS:
Drug: Mirapexin® (Sifrol®)

SUMMARY:
Study to assess the risk of incident heart failure associated with the use of pramipexole compared with other dopamine agonists and additionally, to assess the risk of incident heart failure associated with the use of dopamine agonists in comparison with no use of dopamine agonist therapy

ELIGIBILITY:
Inclusion Criteria:

* All patients between 40 and 89 years of age who received at least one prescription for anti-parkinsonian drugs during the period 1997-2009

Exclusion Criteria:

* Patients with a diagnosis of heart failure or with prescriptions for two or more among the digitalis, angiotensin-converting enzyme (ACE) inhibitors/angiotensin receptor blocker (ARB), and diuretic drug classes prior to cohort entry

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Users of anti-parkinsonian drugs registered with an up-to-standard practice from the United Kingdom's General Practice Research Database (GPRD)
Sampling Method: Non-Probability Sample
Enrollment: 26814 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Assessment of first-time clinical diagnosis of heart failure | 150 months

SECONDARY OUTCOMES:
Overall rate of heart failure | 150 months